CLINICAL TRIAL: NCT03275103
Title: An Open-Label, Multicenter, Phase I Trial Evaluating the Safety and Pharmacokinetics of Escalating Doses of Cevostamab (BFCR4350A) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Dose-Escalation Study of Cevostamab in Participants With Relapsed or Refractory Multiple Myeloma (R/R MM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO39775; 2018-001041-13 (EudraCT Number); 2022-502053-34-00 (Other: EU CT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Arm A: Single Step Dose Escalation for Cevostamab (Experimental): Study drug will be administered intravenously on a 21-day cycle. The step-up dose will be given on Cycle 1 Day 1 and the target dose will be given on C1D8. Subsequently the target dose will be administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Cevostamab
- Arm B: Double Step Dose Escalation for Cevostamab (Experimental): In Cycle 1, participants will receive 2 step-up doses and a target dose. The step-up dose will be given on Cycle 1 Day 1 and C1D8. The target dose will be given on C1D15. Subsequently the target dose will be administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Cevostamab
- Arm C: Single Step Dose Expansion for Cevostamab (Experimental): The single step dose expansion stage of the study may use the dosing and assessment schedule from the single dose escalation arm in Cycle 1, based on data from Arm A.
  Interventions: Drug: Cevostamab
- Arm D: Double Step Dose Expansion for Cevostamab (Experimental): The double step dose expansion stage of the study may use the dosing and assessment schedule from the double step dose escalation arm in Cycle 1, based on data from Arm B.
  Interventions: Drug: Cevostamab
- Arm E: Expansion Phase for Tocilizumab Pretreatment (Experimental): All participants will receive a single dose of tocilizumab intravenously. An additional dose of tocilizumab may be instituted as premedication for subsequent Cycle 1 dose(s) of cevostamab and Cycle 1 cevostamab doses for other treatment arms.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab
- Arm F: Single Step Dose Expansion for Cevostamab (Experimental): The single step dose expansion stage of the study may use the dosing and assessment schedule from the single dose escalation arm in Cycle 1, based on data from Arm A.
  Interventions: Drug: Cevostamab
- Arm G: Double Step Dose Expansion for Cevostamab (Experimental): The double step dose expansion stage of the study may use the dosing and assessment schedule from the double step dose escalation arm in Cycle 1, based on data from Arm B.
  Interventions: Drug: Cevostamab
- Arm H: Triple Step Dose Escalation for Cevostamab (Experimental): In Cycle 1, participants will receive 3 step-up doses and a target dose. The doses will be given on Cycle 1 Days 1, 2-4, 8, and 9-11. Subsequently the target dose will be administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Cevostamab
- Arm I: Triple Step Dose Expansion for Cevostamab (Experimental): The triple step dose expansion stage of the study may use the dosing and assessment schedule from the triple step dose escalation arm in Cycle 1, based on data from Arm H.
  Interventions: Drug: Cevostamab
- Arm J: Expansion Phase for Tocilizumab Pretreatment (Experimental): All participants will receive a single dose of tocilizumab intravenously. An additional dose of tocilizumab may be instituted as premedication for subsequent Cycle 1 dose(s) of cevostamab and Cycle 1 cevostamab doses for other treatment arms.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab
- Arm K: Compressed Double Step Dose Expansion for Cevostamab (Experimental): In Cycle 1, participants will receive 2 step-up doses and a target dose. The doses will be given on Cycle 1 Days 1, 4, and 8. Subsequently the target dose will be administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Cevostamab

INTERVENTIONS:
Drug: Cevostamab — Cevostamab will be administered intravenously on a 21-day cycle, up to a total of 17 cycles.
  Other Names: BFCR4350A; RO7187797
Drug: Tocilizumab — Tocilizumab will be administered as premedication during Cycle 1.
  Other Names: Actemra/RoActemra
  Arms: Arm E: Expansion Phase for Tocilizumab Pretreatment; Arm J: Expansion Phase for Tocilizumab Pretreatment

SUMMARY:
This is a phase I, multicenter, open-label, dose-escalation study of cevostamab administered as a single agent by IV infusion to participants with relapsed or refractory multiple myeloma (R/R MM).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Participants must have relapsed or refractory (R/R) multiple myeloma (MM) for which no established therapy for MM is appropriate and available or be intolerant to those established therapies
* Adverse events from prior anti-cancer therapy resolved to Grade < or = 1, except any grade alopecia and/or peripheral sensory or motor neuropathy which must have resolved to Grade < or = 2
* Measurable disease defined by laboratory test results
* Female participants of childbearing age must agree to remain abstinent or use reliable contraceptive methods during the treatment period, and at least 5 months after last dose of study drug. Women must refrain from breastfeeding during the same period.
* Male participants must agree to refrain from donating sperm, to abstain or use a condom during the treatment period, and for at least 2 months after the last dose of tocilizumab (if applicable).

Exclusion Criteria:

* Inability to comply with protocol-mandated hospitalization and activities restrictions
* Pregnant or breastfeeding, or planning to become pregnant during the study or within 5 months after the last dose of cevostamab or within 3 months after the last dose of of tocilizumab (if applicable)
* Prior use of any monoclonal antibody, radioimmunoconjugate, or antibody-drug conjugate as anti-cancer therapy within 4 weeks before first infusion
* Prior treatment with systemic immunotherapeutic agents within 12 weeks or 5 half-lives of the drug, whichever is shorter, before first infusion
* Prior treatment with chimeric antigen receptor (CAR) T-cell therapy within 12 weeks before first cevostamab infusion
* Known treatment-related, immune-mediated adverse events associated with prior immunotherapeutic agents
* Treatment with radiotherapy, any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first cevostamab infusion
* Autologous stem cell transplantation (SCT) within 100 days prior to first infusion
* Prior allogeneic SCT or solid organ transplantation
* Absolute plasma cell count exceeding 500/micro L or 5% of the peripheral blood white cells
* History of autoimmune disease or of confirmed progressive multifocal leukoencephalopathy
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Patients with known history of amyloidosis (e.g., positive Congo Red stain or equivalent in tissue biopsy)
* Patients with lesions in proximity of vital organs that may develop sudden decompensation/deterioration in the setting of a tumor flare
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Current or past history of central nervous system (CNS) disease, or CNS involvement by MM
* Significant cardiovascular disease that may limit a patient's ability to adequately respond to a CRS event
* Symptomatic active pulmonary disease requiring supplemental oxygen
* Within 14 days prior to first cevostamab infusion: known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics within 4 weeks prior to first infusion
* Positive and quantifiable Epstein-Barr virus (EBV) polymerase chain reaction (PCR) or cytomegalovirus (CMV) PCR prior to first study treatment
* Known or suspected chronic active EBV infection, acute or chronic hepatitis C virus (HCV) infection
* Positive serologic or PCR test results for acute or chronic hepatitis B virus (HBV) infection
* Recent major surgery within 4 weeks prior to first infusion
* Human Immunodeficiency Virus (HIV) positive
* Any episode of active, symptomatic COVID-19 infection, or requiring treatment with IV antivirals for COVID-19 (not including COVID-19 primary prophylaxis) within 14 days, prior to first study treatment
* Administration of a live, attenuated vaccine within 4 weeks before first cevostamab infusion or anticipation that such a live attenuated vaccine will be required during the study
* Received systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents), with the exception of corticosteroid treatment <=10 mg/day prednisone or equivalent within 2 weeks prior to first dose of cevostamab and, if applicable, tocilizumab premedication prior to first dose of cevostamab
* History of illicit drug or alcohol abuse within 12 months prior to screening
* Any medical condition or laboratory test abnormality that precludes the participant's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 8 years
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Up to approximately 8 years
  Dose-Limiting Toxicities (DLTs) will be reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0), except for Cytokine release syndrome (CRS), which will be graded according to the American Society of Transplantation and Cellular Therapy (ASTCT) Consensus Grading for Cytokine Release Syndrome.
Arms E and J Only: Incidence and Severity of Cytokine-release Syndrome (CRS) Following Tocilizumab Premedication Followed by Treatment with Cevostamab | Up to approximately 8 years
  Cytokine release syndrome was recorded as an AE that generally occurs >30 minutes after the start of Cevostamab administration and at any time afterward in a given cycle.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of Cevostamab | Up to approximately 8 years
  Defined as the total exposure of study drug.
AUC of Tocilizumab | Up to approximately 8 years
  Defined as the total exposure of study drug.
Maximum Observed Serum Concentration (Cmax) of Cevostamab | Up to approximately 8 years
  Defined as the maximum observed serum concentration of study drug.
Cmax of Tocilizumab | Up to approximately 8 years
  Defined as the maximum observed serum concentration of study drug.
Minimum Observed Serum Concentration (Cmin) of Cevostamab | Up to approximately 8 years
  Defined as the minimum observed serum concentration of study drug.
Cmin of Tocilizumab | Up to approximately 8 years
  Defined as the minimum observed serum concentration of study drug.
Clearance (CL) of Cevostamab | Up to approximately 8 years
  Defined as the volume of plasma cleared of the drug per unit time.
CL of Tocilizumab | Up to approximately 8 years
  Defined as the volume of plasma cleared of the drug per unit time.
Volume of Distribution at Steady State (Vdss) of Cevostamab | Up to approximately 8 years
  Defined as the actual blood and tissue volume into which a drug is distributed and the relative binding of drug to protein in these spaces.
Vdss of Tocilizumab | Up to approximately 8 years
  Defined as the actual blood and tissue volume into which a drug is distributed and the relative binding of drug to protein in these spaces.
Serum Concentration of Cevostamab | Up to approximately 8 years
Serum Concentration of Tocilizumab | Up to approximately 8 years
Objective Response Rate (ORR) | Up to approximately 8 years
  ORR is defined as percentage of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) .
  sCR is defined as CR (as defined below), plus: Normal FLC ratio and absence of clonal cells in bone marrow (BM) by immunohistochemistry (kappa/lambda ratio </=4:1 or >/=1:2 for kappa and lambda participants, respectively after counting >/=100 plasma cells).
  CR is defined as no evidence of initial monoclonal protein isotype(s) on immunofixation of the serum and urine, disappearance of any soft tissue plasmacytomas, and </= 5% plasma cells in BM.
  VGPR is defined as Serum and urine M-protein detectable by immunofixation but not on electrophoresis; or >/=90% reduction in serum M-protein plus urine M-protein level <100 milligrams (mg)/24 hr.
  PR is defined as >/= 50% reduction of serum M-protein and reduction in 24-hour urine M-protein by >/= 90% or to < 200 mg/24 hours.
Duration of Response | Up to approximately 8 years
  Time from first occurrence of ORR (defined previously) to disease progression (PD) or death from any cause. PD: increase of >/=25% from lowest response value in one of the following: serum M-protein (absolute increase >/=0.5 grams per deciliter (g/dL); serum M-protein increase >/=1g/dL, if lowest M component was >/=5g/dL; urine M-protein (absolute increase >/=200 mg/24 hours); no measurable serum and urine M-protein levels: difference between involved and uninvolved free light chain (FLC) levels (absolute increase >10 mg/dL); no measurable serum and urine M-protein levels and no measurable disease by FLC: BM plasma cell % irrespective of baseline status (absolute % >/=10%); new lesion(s) >/=50% increase from lowest point in sum of the products of diameters of > 1 lesion, or >/=50% increase in longest diameter of a previous lesion >1 centimeter (cm) in short axis; >/=50% increase in circulating plasma cells (minimum 200 cells per microliter) if only measure of disease.
Change from Baseline in the Presence Anti-Drug Antibodies (ADAs) | Up to approximately 8 years
  To evaluate the immune response to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (17):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital - Arizona, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of Colorado Denver, Aurora, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Peter MacCallum Cancer Center, East Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Canada (3):
  - University of Calgary Cumming School of Medicine, Calgary, Alberta
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona/iruña, Navarre
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No